CLINICAL TRIAL: NCT03267329
Title: A Randomized, Open, Parallel, Multicenter, Phase 4 Study to Evaluate the Central Aortic Pressure Effect Between Fixed Dose Combination (Duowell® Tab) and Monotherapy of Telmisartan in Mild Dyslipidemia Patients With Hypertension
Brief Title: Duowell® vs. Telmisartan Monotherapy in Mild Dyslipidemia Patients With Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMC023
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2020-05

CONDITIONS: Hypertension; Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — Telmisartan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duowell® Tab. (Experimental): Once daily during 16 wks
  Interventions: Drug: Duowell®
- Telmisartan (Active Comparator): Once daily during 16 wks
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Duowell® — telmisartan 80mg/rosuvastatin 10mg for ASCVD risk=5%~7.5% or telmisartan 80mg/rosuvastatin 20mg for ASCVD risk≥7.5%
  Arms: Duowell® Tab.
Drug: Telmisartan — telmisartan 80mg
  Arms: Telmisartan

SUMMARY:
This study is to evaluate effect and safety on central blood pressure with Duowell compared to telmisartan monotherapy in mild dyslipidemia patients with hypertension during 16 weeks.

ELIGIBILITY:
Inclusion Criteria (All of the followings)

* 40 to 75 years old diagnosed with hypertension
* at screening, SBP ≥ 140 mmHg
* at randomization, 130 mmHg ≤ SBP ≤160 mmHg or 80 mmHg ≤ DBP ≤ 100 mmHg
* at screening, ASCVD risk ≥ 5 %
* Those who did not take the dyslipidemic medications during screening or who stopped medication for more than 2 months
* at screening, 130 mg/dL ≤ Calculated (or Measured) Serum LDL-C ≤ 190 mg/dL
* Pregnancy test negative and and who has agreed to perform effective contraception during the clinical trial

Exclusion Criteria (Any of the followings)

* known hypersensitivity to AT-1 receptor blockers or statins
* Those who are treated with secondary hypertension during screening
* Those who are being treated for malignant hypertension during screening
* Those who are taking concurrent medication that may affect blood pressure during screening
* Those who have been diagnosed with myocardial infarction or unstable angina or stroke within the last 6 months at screening
* Patients with heart failure NYHA III-IV or Left Ventricular Ejection Fraction <40% within the last 6 months at screening
* Patients with valve disease with hemodynamically significant (over moderate degree) obstructive
* Those with known atrial fibrillation or atrioventricular conduction disturbance
* Those who show the following numerical values during the screening test

  1. CPK ≥ 3 times the normal upper limit
  2. Serum Creatinine > 3 mg/dL
  3. Serum Potassium > 5.5 mmol/L
  4. ALT or AST ≥ 3 times the upper normal limit
* Those with known bilateral renal artery stenosis
* Patients who underwent open heart surgery within 4 weeks prior to randomization and who had a cardiac surgery plan
* Those taking statins within 8 weeks before randomization
* Those with severe obstructive, limited or other pulmonary disease history
* Those with non-cardiac disease that can significantly shorten the expected life span to less than 2 years (eg, severe cancer)
* at screening, Anti-HIV Ab, HBsAg, HCV Ab positive

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in mean central systolic blood pressure | at week 16

SECONDARY OUTCOMES:
Changes from baseline in mean brachial systolic blood pressure | at week 4 and at week 16 and at week 28
Changes from baseline in mean brachial pulse pressure | at week 4 and at week 16 and and at week 28
Changes from mean brachial diastolic blood pressure | at week 4 and at week 16 and at week 28
Changes from baseline in augmentation index | at week 16 and at week 28
Changes from baseline in carotid femoral pulse wave velocity | at week 16 and at week 28

OTHER OUTCOMES:
Changes from baseline in central blood pressure according to the frequency of access in mobile application | up to 4 weeks and up to 16 weeks
Drug compliance between over 50% and less 50% of assessment in mobile application | at week 4 weeks and at week 16
Drug compliance between over 50% and less 50% of assessment in mobile application | up to 3 months end of study
Changes from the end of treatment in central systolic blood pressure after 3 months | at 3 months from the end of study
Numbers of inconvenience reported by mobile application at each visit | up to 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No